CLINICAL TRIAL: NCT02622295
Title: Musculoskeletal Plasticity After Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Richard K Shields (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Richard K Shields, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 200412709; R01HD084645 (NIH)
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Results first posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-08

CONDITIONS: Spinal Cord Injuries
Keywords: metabolism; glucose; osteoporosis; secondary health conditions; quality of life; standing; electrical stimulation; diabetes; insulin; skeletal muscle
MeSH Terms: conditions — Spinal Cord Injuries; Osteoporosis; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acute gene regulation (Experimental): Adaptations in gene regulation in response to single-session electrically induced exercise
  Interventions: Behavioral: Single-session electrically induced exercise
- Training Study (Experimental): Adaptations in gene regulation, metabolic markers, and subject-report metrics in response to up to 3 years of electrically induced exercise
  Interventions: Behavioral: Electrically-induced exercise training

INTERVENTIONS:
Behavioral: Single-session electrically induced exercise — A single session of electrically induced exercise to the quadriceps and hamstring muscle groups of people with paralysis.
  Arms: Acute gene regulation
Behavioral: Electrically-induced exercise training — Multiple sessions of electrically induced exercise to the quadriceps and hamstring muscle groups for up to 3 years in people with paralysis.
  Arms: Training Study

SUMMARY:
Patients with spinal cord injury (SCI) experience metabolic syndrome, diabetes, obesity, pressure ulcers, and cardiovascular disease at far greater rates than the general population. A rehabilitation method to prevent or reverse the systemic metabolic consequences of SCI is a pressing need. The purpose of this study is to determine the dose of muscle activity that can enhance an oxidative muscle phenotype and improve clinical markers of metabolic health and bone turnover in patients with SCI. The long-term goal of this research is to develop exercise-based interventions to prevent secondary health conditions such as diabetes and to ultimately protect health-related quality of life (QOL). Specific Aim 1: To compare changes in skeletal muscle gene regulation in individuals who receive high frequency (HF) active-resisted stance and low frequency (LF) active-resisted stance for 3 years. Hypothesis 1: The expression of genes regulating skeletal muscle metabolism will support that HF and LF both instigate a shift toward an oxidative muscle phenotype. A novel finding will be that LF is a powerful regulator of oxidative pathways in skeletal muscle. Specific Aim 2: To compare changes in systemic markers of metabolic health and bone turnover in individuals with SCI who receive HF or LF for 3 years. Hypothesis 2: HF and LF will both reduce glucose/insulin levels and HOMA (homeostasis model assessment) score.

Secondary Aim: To measure subject-reported QOL using the EQ-5D survey metric. Hypothesis 3: HF and LF subjects will show a trend toward improved self-reported QOL after 3 years. There will be an association between metabolic improvement and improved perception of QOL. These observations will support that this intervention has strong feasibility for future clinical translation.

ELIGIBILITY:
Inclusion Criteria:

* Motor complete SCI (AIS A-B)

Exclusion Criteria:

1. Pressure ulcers
2. Chronic infection
3. Lower extremity muscle contractures
4. Deep vein thrombosis
5. Bleeding disorder
6. Recent limb fractures
7. Any comorbid disease known to affect bone metabolism (such as parathyroid dysfunction)
8. Pregnancy
9. Anti-osteoporosis medications
10. Vitamin D supplements
11. Metformin or other medications for diabetes.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Shields, PhD, PT, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dudley-Javoroski S, Saha PK, Liang G, Li C, Gao Z, Shields RK. High dose compressive loads attenuate bone mineral loss in humans with spinal cord injury. Osteoporos Int. 2012 Sep;23(9):2335-46. doi: 10.1007/s00198-011-1879-4. Epub 2011 Dec 21. PMID 22187008
- [Background] Dudley-Javoroski S, Shields RK. Dose estimation and surveillance of mechanical loading interventions for bone loss after spinal cord injury. Phys Ther. 2008 Mar;88(3):387-96. doi: 10.2522/ptj.20070224. Epub 2008 Jan 17. PMID 18202080
- [Background] Dudley-Javoroski S, Shields RK. Active-resisted stance modulates regional bone mineral density in humans with spinal cord injury. J Spinal Cord Med. 2013 May;36(3):191-9. doi: 10.1179/2045772313Y.0000000092. PMID 23809588
- [Background] Dudley-Javoroski S, Littmann AE, Iguchi M, Shields RK. Doublet stimulation protocol to minimize musculoskeletal stress during paralyzed quadriceps muscle testing. J Appl Physiol (1985). 2008 Jun;104(6):1574-82. doi: 10.1152/japplphysiol.00892.2007. Epub 2008 Apr 24. PMID 18436697
- [Background] Dudley-Javoroski S, Shields RK. Assessment of physical function and secondary complications after complete spinal cord injury. Disabil Rehabil. 2006 Jan 30;28(2):103-10. doi: 10.1080/09638280500163828. PMID 16393840
- [Background] Adams CM, Suneja M, Dudley-Javoroski S, Shields RK. Altered mRNA expression after long-term soleus electrical stimulation training in humans with paralysis. Muscle Nerve. 2011 Jan;43(1):65-75. doi: 10.1002/mus.21831. PMID 21171097
- [Background] Frey Law LA, Shields RK. Femoral loads during passive, active, and active-resistive stance after spinal cord injury: a mathematical model. Clin Biomech (Bristol). 2004 Mar;19(3):313-21. doi: 10.1016/j.clinbiomech.2003.12.005. PMID 15003348
- [Background] Kunkel SD, Suneja M, Ebert SM, Bongers KS, Fox DK, Malmberg SE, Alipour F, Shields RK, Adams CM. mRNA expression signatures of human skeletal muscle atrophy identify a natural compound that increases muscle mass. Cell Metab. 2011 Jun 8;13(6):627-38. doi: 10.1016/j.cmet.2011.03.020. PMID 21641545
- [Background] McHenry CL, Wu J, Shields RK. Potential regenerative rehabilitation technology: implications of mechanical stimuli to tissue health. BMC Res Notes. 2014 Jun 3;7:334. doi: 10.1186/1756-0500-7-334. PMID 24894666
- [Background] McHenry CL, Shields RK. A biomechanical analysis of exercise in standing, supine, and seated positions: Implications for individuals with spinal cord injury. J Spinal Cord Med. 2012 May;35(3):140-7. doi: 10.1179/2045772312Y.0000000011. PMID 22507023
- [Background] Petrie MA, Suneja M, Faidley E, Shields RK. A minimal dose of electrically induced muscle activity regulates distinct gene signaling pathways in humans with spinal cord injury. PLoS One. 2014 Dec 22;9(12):e115791. doi: 10.1371/journal.pone.0115791. eCollection 2014. PMID 25531450
- [Background] Petrie MA, Suneja M, Faidley E, Shields RK. Low force contractions induce fatigue consistent with muscle mRNA expression in people with spinal cord injury. Physiol Rep. 2014 Feb 25;2(2):e00248. doi: 10.1002/phy2.248. eCollection 2014 Feb 1. PMID 24744911
- [Background] Shields RK, Dudley-Javoroski S. Monitoring standing wheelchair use after spinal cord injury: a case report. Disabil Rehabil. 2005 Feb 4;27(3):142-6. doi: 10.1080/09638280400009337. PMID 15823996
- [Background] Petrie M, Suneja M, Shields RK. Low-frequency stimulation regulates metabolic gene expression in paralyzed muscle. J Appl Physiol (1985). 2015 Mar 15;118(6):723-31. doi: 10.1152/japplphysiol.00628.2014. Epub 2015 Jan 29. PMID 25635001
- [Background] Zhorne R, Dudley-Javoroski S, Shields RK. Skeletal muscle activity and CNS neuro-plasticity. Neural Regen Res. 2016 Jan;11(1):69-70. doi: 10.4103/1673-5374.169623. No abstract available. PMID 26981083
- [Background] Petrie MA, Kimball AL, McHenry CL, Suneja M, Yen CL, Sharma A, Shields RK. Distinct Skeletal Muscle Gene Regulation from Active Contraction, Passive Vibration, and Whole Body Heat Stress in Humans. PLoS One. 2016 Aug 3;11(8):e0160594. doi: 10.1371/journal.pone.0160594. eCollection 2016. PMID 27486743
- [Background] Shields RK. Turning Over the Hourglass. Phys Ther. 2017 Oct 1;97(10):949-963. doi: 10.1093/ptj/pzx072. PMID 29029555
- [Background] Woelfel JR, Kimball AL, Yen CL, Shields RK. Low-Force Muscle Activity Regulates Energy Expenditure after Spinal Cord Injury. Med Sci Sports Exerc. 2017 May;49(5):870-878. doi: 10.1249/MSS.0000000000001187. PMID 28009786
- [Background] Yen CL, McHenry CL, Petrie MA, Dudley-Javoroski S, Shields RK. Vibration training after chronic spinal cord injury: Evidence for persistent segmental plasticity. Neurosci Lett. 2017 Apr 24;647:129-132. doi: 10.1016/j.neulet.2017.03.019. Epub 2017 Mar 16. PMID 28315725
- [Background] Oza PD, Dudley-Javoroski S, Shields RK. Modulation of H-Reflex Depression with Paired-Pulse Stimulation in Healthy Active Humans. Rehabil Res Pract. 2017;2017:5107097. doi: 10.1155/2017/5107097. Epub 2017 Oct 31. PMID 29225972
- [Background] Woelfel JR, Dudley-Javoroski S, Shields RK. Precision Physical Therapy: Exercise, the Epigenome, and the Heritability of Environmentally Modified Traits. Phys Ther. 2018 Nov 1;98(11):946-952. doi: 10.1093/ptj/pzy092. PMID 30388254
- [Background] Cole KR, Dudley-Javoroski S, Shields RK. Hybrid stimulation enhances torque as a function of muscle fusion in human paralyzed and non-paralyzed skeletal muscle. J Spinal Cord Med. 2019 Sep;42(5):562-570. doi: 10.1080/10790268.2018.1485312. Epub 2018 Jun 20. PMID 29923814
- [Background] Dudley-Javoroski S, Lee J, Shields RK. Cognitive function, quality of life, and aging: relationships in individuals with and without spinal cord injury. Physiother Theory Pract. 2022 Jan;38(1):36-45. doi: 10.1080/09593985.2020.1712755. Epub 2020 Jan 8. PMID 31914347
- [Background] Petrie MA, Sharma A, Taylor EB, Suneja M, Shields RK. Impact of short- and long-term electrically induced muscle exercise on gene signaling pathways, gene expression, and PGC1a methylation in men with spinal cord injury. Physiol Genomics. 2020 Feb 1;52(2):71-80. doi: 10.1152/physiolgenomics.00064.2019. Epub 2019 Dec 23. PMID 31869286
- [Background] Lee J, Dudley-Javoroski S, Shields RK. Motor demands of cognitive testing may artificially reduce executive function scores in individuals with spinal cord injury. J Spinal Cord Med. 2021 Mar;44(2):253-261. doi: 10.1080/10790268.2019.1597482. Epub 2019 Apr 3. PMID 30943119
- [Background] Shields RK. Precision Rehabilitation: How Lifelong Healthy Behaviors Modulate Biology, Determine Health, and Affect Populations. Phys Ther. 2022 Jan 1;102(1):pzab248. doi: 10.1093/ptj/pzab248. No abstract available. PMID 34718793
- [Background] Shields RK, Dudley-Javoroski S. Epigenetics and the International Classification of Functioning, Disability and Health Model: Bridging Nature, Nurture, and Patient-Centered Population Health. Phys Ther. 2022 Jan 1;102(1):pzab247. doi: 10.1093/ptj/pzab247. PMID 34718813
- [Background] Petrie MA, Taylor EB, Suneja M, Shields RK. Genomic and Epigenomic Evaluation of Electrically Induced Exercise in People With Spinal Cord Injury: Application to Precision Rehabilitation. Phys Ther. 2022 Jan 1;102(1):pzab243. doi: 10.1093/ptj/pzab243. PMID 34718779

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acute Gene Regulation | Training Study
Started | 40 | 31
Completed | 40 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acute Gene Regulation | Training Study | Total
Number analyzed (Participants) | 40 | 31 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 31 | 71
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 27 | 21 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 39 | 31 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 34 | 28 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 31 | 71
Quadriplegia versus Paraplegia [Count of Participants; unit: Participants]
  Quadriplegia | 14 | 11 | 25
  Paraplegia | 26 | 20 | 46

OUTCOME MEASURES:

1. Primary Outcome: Acute Gene Regulation: MSTN
Description: Acute post-stimulation effect upon skeletal muscle myostatin (MSTN) expression, measured via muscle biopsy and exon array analysis. Probe summarization and probe set normalization were performed using robust multichip average, which included background correction, quantile normalization, log2 transformation and median polish probe set summarization. 0 represents no mRNA expression and higher values represent greater expression compared to all genes in the microarray.
Time Frame: 3 hours after a single session of electrical stimulation
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Acute Gene Regulation
Number analyzed (Participants) | 40
arbitrary units
  Pre-Stimulation | 5.49 (0.633)
  Post-Stimulation | 4.76 (0.748)
Statistical Analysis 1: Comparison: Acute Gene Regulation; Test type: Superiority; p < 0.001, ANOVA

2. Primary Outcome: Acute Gene Regulation: PGC1-alpha
Description: Acute post-stimulation effect upon skeletal muscle peroxisome proliferator-activated receptor gamma coactivator alpha (PGC1-alpha) expression, measured via muscle biopsy and exon array analysis. Probe summarization and probe set normalization were performed using robust multichip average, which included background correction, quantile normalization, log2 transformation and median polish probe set summarization. 0 represents no mRNA expression and higher values represent greater expression compared to all genes in the microarray.
Time Frame: 3 hours after a single session of electrical stimulation
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Acute Gene Regulation
Number analyzed (Participants) | 40
arbitrary units
  Pre-Stimulation | 5.23 (0.486)
  Post-Stimulation | 6.63 (0.395)
Statistical Analysis 1: Comparison: Acute Gene Regulation; Test type: Superiority; p < 0.001, ANOVA

3. Primary Outcome: Acute Gene Regulation: PDK4
Description: Acute post-stimulation effect upon skeletal muscle pyruvate dehydrogenase kinase, isozyme 4 (PDK4-alpha) expression, measured via muscle biopsy and exon array analysis. Probe summarization and probe set normalization were performed using robust multichip average, which included background correction, quantile normalization, log2 transformation and median polish probe set summarization. 0 represents no mRNA expression and higher values represent greater expression compared to all genes in the microarray.
Time Frame: 3 hours after a single session of electrical stimulation
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Acute Gene Regulation
Number analyzed (Participants) | 40
arbitrary units
  Pre-Stimulation | 6.59 (0.413)
  Post-Stimulation | 7.29 (0.416)
Statistical Analysis 1: Comparison: Acute Gene Regulation; Test type: Superiority; p < 0.001, ANOVA

4. Primary Outcome: Acute Gene Regulation: SDHB
Description: Acute post-stimulation effect upon skeletal muscle succinate dehydrogenase-B (SDHB) expression, measured via muscle biopsy and exon array analysis. Probe summarization and probe set normalization were performed using robust multichip average, which included background correction, quantile normalization, log2 transformation and median polish probe set summarization. 0 represents no mRNA expression and higher values represent greater expression compared to all genes in the microarray.
Time Frame: 3 hours after a single session of electrical stimulation
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Acute Gene Regulation
Number analyzed (Participants) | 40
arbitrary units
  Pre-Stimulation | 7.15 (0.478)
  Post-Stimulation | 7.20 (0.490)
Statistical Analysis 1: Comparison: Acute Gene Regulation; Test type: Superiority; p = 0.467, ANOVA

5. Primary Outcome: Post-training Gene Regulation: MSTN
Description: Pre- and post-training skeletal muscle myostatin (MSTN) expression, measured via muscle biopsy and exon array analysis. Probe summarization and probe set normalization were performed using robust multichip average, which included background correction, quantile normalization, log2 transformation and median polish probe set summarization. 0 represents no mRNA expression and higher values represent greater expression compared to all genes in the microarray.
Time Frame: up to 3 years
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Training Study
Number analyzed (Participants) | 31
arbitrary units
  Baseline | 5.34 (0.510)
  Post-Training (up to 3 years) | 4.78 (0.668)
Statistical Analysis 1: Comparison: Training Study; Test type: Superiority; p < 0.001, ANOVA

6. Primary Outcome: Post-training Gene Regulation: PGC1-alpha
Description: Pre- and post-training skeletal muscle peroxisome proliferator-activated receptor gamma coactivator alpha (PGC1-alpha) expression, measured via muscle biopsy and exon array analysis. Probe summarization and probe set normalization were performed using robust multichip average, which included background correction, quantile normalization, log2 transformation and median polish probe set summarization. 0 represents no mRNA expression and higher values represent greater expression compared to all genes in the microarray.
Time Frame: up to 3 years
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Training Study
Number analyzed (Participants) | 31
arbitrary units
  Baseline | 5.89 (0.372)
  Post-Training (up to 3 years) | 5.90 (0.337)
Statistical Analysis 1: Comparison: Training Study; Test type: Superiority; p = 0.932, ANOVA

7. Primary Outcome: Post-training Gene Regulation: PDK4
Description: Pre- and post-training skeletal muscle pyruvate dehydrogenase kinase, isozyme 4 (PDK4-alpha) expression, measured via muscle biopsy and exon array analysis. Probe summarization and probe set normalization were performed using robust multichip average, which included background correction, quantile normalization, log2 transformation and median polish probe set summarization. 0 represents no mRNA expression and higher values represent greater expression compared to all genes in the microarray.
Time Frame: up to 3 years
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Training Study
Number analyzed (Participants) | 31
arbitrary units
  Baseline | 7.01 (0.377)
  Post-Training (up to 3 years) | 6.87 (0.372)
Statistical Analysis 1: Comparison: Training Study; Test type: Superiority; p = 0.326, ANOVA

8. Primary Outcome: Post-training Gene Regulation: SDHB
Description: Pre- and post-training skeletal muscle succinate dehydrogenase-B (SDHB) expression, measured via muscle biopsy and exon array analysis. Probe summarization and probe set normalization were performed using robust multichip average, which included background correction, quantile normalization, log2 transformation and median polish probe set summarization. 0 represents no mRNA expression and higher values represent greater expression compared to all genes in the microarray.
Time Frame: up to 3 years
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Training Study
Number analyzed (Participants) | 31
arbitrary units
  Baseline | 7.22 (0.456)
  Post-Training (up to 3 years) | 7.26 (0.556)
Statistical Analysis 1: Comparison: Training Study; Test type: Superiority; p = 0.673, ANOVA

9. Primary Outcome: Post-training Metabolism: Fasting Glucose
Description: Pre- and post-training fasting glucose, measured via venipuncture and standard laboratory assays
Time Frame: up to 3 years
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Training Study
Number analyzed (Participants) | 10
mg/dL
  Baseline | 95.5 (10.5)
  Post-Training (up to 3 years) | 97.8 (7.7)
Statistical Analysis 1: Comparison: Training Study; Test type: Superiority; p = 0.539, ANOVA

10. Primary Outcome: Post-training Metabolism: Fasting Insulin
Description: Pre- and post-training fasting insulin, measured via venipuncture and standard laboratory assays
Time Frame: up to 3 years
Measure: Mean (Standard Deviation); unit: microU/mL
Arm/Group | Training Study
Number analyzed (Participants) | 10
microU/mL
  Baseline | 20.6 (16.7)
  Post-Training (up to 3 years) | 11.8 (8.37)
Statistical Analysis 1: Comparison: Training Study; Test type: Superiority; p = 0.155, ANOVA

11. Primary Outcome: Post-training Metabolism: HOMA Score
Description: Pre- and post-training HOMA score, calculated via the Homeostasis Model Assessment equation.
  Maximum/minimum values: not applicable. Scores >2 are indicative of insulin resistance.
Time Frame: up to 3 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Training Study
Number analyzed (Participants) | 10
score on a scale
  Baseline | 2.3 (1.8)
  Post-Training (up to 3 years) | 1.3 (0.9)
Statistical Analysis 1: Comparison: Training Study; Test type: Superiority; p = 0.164, ANOVA

12. Primary Outcome: Post-training Bone Turnover: Osteocalcin
Description: Pre- and post-training serum osteocalcin, measured via venipuncture and enzyme-linked immunosorbent assay
Time Frame: up to 3 years
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Training Study
Number analyzed (Participants) | 10
pg/mL
  Baseline | 6638.5 (2711.9)
  Post-Training (up to 3 years) | 6874.1 (3197.5)
Statistical Analysis 1: Comparison: Training Study; Test type: Superiority; p = 0.493, ANOVA

13. Secondary Outcome: Post-training Subject-report Measures: EQ-5D
Description: Pre- and post-training QALY (quality-adjusted life-years) via the EQ-5D subject-report survey instrument.
  Scale ranges from -0.287 to 0.992. Higher values indicated a higher self-perceived health state.
Time Frame: up to 3 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Training Study
Number analyzed (Participants) | 11
score on a scale
  Baseline | 0.296 (0.111)
  Post-Training (up to 3 years) | 0.265 (0.093)
Statistical Analysis 1: Comparison: Training Study; Test type: Superiority; p = 0.458, ANOVA

ADVERSE EVENTS:
Time Frame: From Baseline up to 3 years
Arm/Group | Acute Gene Regulation | Training Study
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/31
Other Adverse Events (participants affected / at risk) | 0/40 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT02622295/Prot_SAP_000.pdf